CLINICAL TRIAL: NCT07074067
Title: V-Notes Hysterectomy in Patients With Endometrial cáncer Compared With Laparoscopic Surgery (Robotically Assisted or Not): ENOLA TRIAL
Acronym: ENOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4-5-HCUVA
Record Dates: First submitted 2025-06-27; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Adenocarcinoma
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: prospective, open-label, longitudinal, randomized, longitudinal, blind-blind third-party (observer-blind)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic surgery (Active Comparator): within the laparoscopic (LPC) arm, 21 patients will be assigned to conventional LPC and another 21 to robotic surgery, consecutively.
  Interventions: Procedure: Laparoscopic surgery
- surgery via v-NOTES (Experimental): surgery via v-NOTES
  Interventions: Procedure: surgery via v-NOTES

INTERVENTIONS:
Procedure: Laparoscopic surgery — the laparoscopic (LPC) arm, 21 patients will be assigned to conventional LPC and another 21 to robotic surgery, consecutively.
  Arms: Laparoscopic surgery
Procedure: surgery via v-NOTES — surgery via v-NOTES
  Arms: surgery via v-NOTES

SUMMARY:
The v-NOTES surgical approach may provide important advantages over the already established effective technique (laparoscopy) for safely and successfully removing the uterus and adnexa in patients with low-grade endometrioid adenocarcinoma FIGO IA and atypical endometrial hyperplasia, such as a better aesthetic outcome, a shorter hospital stays, and a decrease in pain and postoperative complications. without increasing surgical time and with equal safety for the patient.

DETAILED DESCRIPTION:
A prospective, open-label, longitudinal, randomized, longitudinal, blind-blind third-party (observer-blind) clinical trial will be conducted. Patients with a diagnosis of endometrioid adenocarcinoma IA G1-G2 and atypical endometrial hyperplasia will be recruited in the Gynecology Oncology consultations of the HCUVA. Patients who meet all the inclusion criteria and none of the exclusion criteria from the trial will be informed about the study, and if they agree to participate, they will sign the informed consent. The data will be included in the Hospital's computer system (Selene), and will be compiled in a database that will be accessible only by the physicians included in the study. Subsequently, this database will be analysed by a statistician from outside the HCUVA's Gynaecology Service. After surgery, patients will be monitored after surgery, first on the hospitalization floor prior to discharge, and later in face-to-face consultations as well as by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Age of majority (> 18 years)
* Willingness to participate in the study and signing of informed consent
* Histological diagnosis, by endometrial biopsy (either using a Cornier cannula or directed by diagnostic hysteroscopy) of atypical endometrial hyperplasia or low-grade endometrioid adenocarcinoma (G1-G2), with an initial stage (IA) at preoperative evaluation

Exclusion Criteria:

Pregnant Women

* Nullicottitis
* Severe uterine prolapse (grade IV)
* Large myomatous uterus (greater than 18 weeks of gestation)
* Severe comorbidities that contraindicate surgery, such as sepsis, severe renal failure, severe cardiopulmonary disease, or severe coagulopathies 33
* Presence of previous illnesses or treatments that may have caused severe pelvic adhesions that obliterate the Douglas pouch and prevent vaginal entry, such as deep pelvic endometriosis, severe pelvic inflammatory disease, inflammatory bowel disease (ulcerative colitis, diverticulitis, Crohn's disease), or a history of pelvic radiotherapy, among others
* Concomitant presence of adnexal masses or formations of considerable size that are expected to substantially lengthen the uterus Surgical time due to the difficulty of extraction
* Contraindication to general anesthesia
* Active pelvic or lower urinary tract infection
* Clinical suspicion of advanced stage of the neoplasia
* Any histological type of endometrial cancer other than those described previously.
* High histological grade (G3)
* Current abnormality in cervical cytology (CVC) requiring more aggressive surgical intervention
* Revocation of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with endometrial cancer
Enrollment: 84 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Time taken to perform surgery | Perioperative
  Surgical time will be defined, in the case of the laparoscopic/robotic route, as the time elapsed from the insertion of the first trocar to the removal of the last one, and in the case of the v-NOTES route, as the time elapsed from the beginning of the vaginal surgery to the end of the surgery. The previous time of positioning of the patient, anesthesia, asepsis and sizing of the surgical field will not be taken into account

SECONDARY OUTCOMES:
AGE | Day 1
  Number of years
Body Mass Index | Day 1
  numerical variable measured in "Kg/m2
times spent in surgical techniques | 1 day post surgery
  number of minutes the surgery lasts
Measurement of post-surgical pain | 6 and 24 hours after the intervention
  using the Visual Analog Scale (VAS) in the immediate postoperative period It consists of a 10-centimeter straight line, where one end represents the absence of pain (0) and the other, the worst pain imaginable (10).
Study of overall patient satisfaction upon hospital discharge | Trough study completion, an average of a1 year
  Study of overall patient satisfaction upon hospital discharge: "SERVQHOS (quality of hospital services) a questionnaire to assess the perceived quality of hospital care through 20 items across 5 dimensions, each item is rated using a Likert-type(1-7) scale allowing free subjective evaluation.
Study of patient quality of life before and one month after surgery | 0, 30 days post surgery
  SF12 V2 Quality of Life Questionnaire"SF-12v2 is a shortened form (12 items) of the SF-36v2 Health Survey. (minimum 20 points maximum 60 points)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Guijarro Campillo, MD, Principal Investigator — HCUVA
Locations (1):
- HCUVA, Murcia, Murcia, Spain